CLINICAL TRIAL: NCT06140069
Title: Voluntary Termination of Pregnancy Between 14 and 16 Weeks of Amenorrhea: Comparison of Women's Experiences Depending on the Method Used, Surgical or Medicinal.
Brief Title: Voluntary Termination of Pregnancy: Comparison of Women's Experiences Depending on the Method Used.
Acronym: VECUVG
Status: Withdrawn | Type: Observational
Why Stopped: too few patients undergoing medical abortion (< 5 per year)
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0563
Record Dates: First submitted 2023-11-10; First posted 2023-11-18 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Voluntary Termination of Pregnancy
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Experimental: Patient treated at the Toulouse University Hospital for an abortion: Patient treated at the Toulouse University Hospital for an abortion between 14 and 16 weeks (dating by ultrasound) presenting with a single and evolving pregnancy.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A questionnaire is offered to patients who meet the eligibility criteria and who have given their non-objection during the abortion request consultation.
  This questionnaire includes questions for screening for anxiety and depressive disorders.

SUMMARY:
Voluntary termination of pregnancy (abortion) is a major current societal issue. This is a very common situation, around 225,000 abortions are carried out every year in France. The French law of March 2, 2022 (no. 2022-295) extended the legal deadline for voluntary termination of pregnancy from 14 to 16 weeks of amenorrhea (SA). The recommendations have not been updated following this legal extension, the centers performing abortions are therefore free regarding the protocol for carrying out these so-called late abortions (between 14 and 16 weeks). There are two pregnancy termination techniques practiced in France: medical or surgical. The drug method consists of drug-induced expulsion of the pregnancy. This method is carried out in the delivery room, and lasts several hours. The surgical method consists of an endouterine aspiration carried out in the operating room, which lasts approximately 30 minutes. At the Toulouse University Hospital, as in many centers in France, it is the patient who chooses the method, apart from a contraindication to one or other of these methods. Due to the recent nature of these late abortions, practitioners still have little experience of the consequences of these procedures and this compromises the quality of the information provided to patients. It is necessary to have quality studies to improve knowledge about late abortions, in order to be able to correctly inform patients and allow them to make an informed choice regarding the method used.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient
* Having given her non-opposition after clear and fair information (patient who understands and reads French)
* Patient treated at the Toulouse University Hospital for an abortion between 14 and 16 weeks (dating by ultrasound)
* Singleton pregnancy
* Progressive pregnancy

Exclusion Criteria:

* Protected adult patient (guardianship, curatorship, protection of justice)
* Developing psychiatric pathologies
* Fetal anomaly detected

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient coming for Voluntary termination of pregnancy (abortion)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of anxiety or depressive disorder depending on the method used, surgical or medicinal | At the inclusion visit before abortion and 3 weeks after abortion
  Anxiety will be measured using Hospital Anxiety and Depression Scale (HADS)

CONTACTS AND LOCATIONS:
Overall Officials: Lola LOUSSERT CHAMBRE, MD, Principal Investigator — University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No